CLINICAL TRIAL: NCT03027609
Title: Placebo-controlled, Double-blind, Randomized Study of Aerucin® as Adjunct Therapy to Antibiotics in the Treatment of P. Aeruginosa Pneumonia
Brief Title: Adjunctive Therapeutic Treatment With Human Monoclonal Antibody AR-105 (Aerucin®) in P. Aeruginosa Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-105-002
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2019-08

CONDITIONS: Pseudomonas Aeruginosa Pneumonia
Keywords: Pseudomonas aeruginosa; pneumonia
MeSH Terms: conditions — Pseudomonas Infections; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR-105 (Experimental): One intravenous infusion of AR-105 20mg/'kg
  Interventions: Drug: AR-105
- Control (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR-105 — monoclonal antibody
  Other Names: Aerubumab; Aerucin
  Arms: AR-105
Drug: Placebo — matching placebo (+ SOC antibiotics)
  Other Names: Control (SOC antibiotics)
  Arms: Control

SUMMARY:
Prospective, double-blind, randomized assessment of the efficacy, safety and pharmacokinetic of Aerucin® as adjunct treatment (in addition to standard of care antibiotics) for pneumonia caused by P. aeruginosa.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study of the human monoclonal antibody (mAb) AR-105 for the adjunctive therapeutic treatment of P. aeruginosa pneumonia in mechanically ventilated subjects. Subjects who are randomized will be treated with either standard of care (SOC) antibiotics plus placebo or SOC antibiotics plus AR-105. The study is being conducted at approximately 100 clinical sites across 17 countries. Subjects who meet all of the inclusion criteria and none of the exclusion criteria are screened by the microbiological culture test and/or rapid diagnostic test of an endotracheal aspirate to confirm the presence of an active P. aeruginosa infection. Following eligibility confirmation, the subject will be randomized in a 1:1 ratio to one of two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* ≥18 years of age, ≥ 20 years of age (Taiwan only),≥ 19 (S. Korea only)
* pneumonia due to P. aeruginosa
* mechanically-ventilated
* intubated
* APACHE II score between 10 and 35

Exclusion Criteria (main criteria):

* being moribund
* effective antibiotic therapy ≥48 hours
* immunocompromised
* underlying pulmonary disease that may preclude the assessment of a therapeutic response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (105):
- United States (14):
  - Research Site 1, Sacramento, California
  - Research Site 2, San Diego, California
  - Research Site 3, Jacksonville, Florida
  - Research Site 4, Tampa, Florida
  - Research Site 5, Chicago, Illinois
  - Research Site 6, Lexington, Kentucky
  - Research Site 7, Detroit, Michigan
  - Research Site 8, Detroit, Michigan
  - Research Site 9, Royal Oak, Michigan
  - Research Site 10, St Louis, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
- Australia (2):
  - Research Site, Adelaide
  - Research Site, Woolloongabba
- Belarus (5):
  - Research Site, Brest
  - Research Site, Grodno
  - Research Site, Homyel
  - Research Site, Minsk
  - Research Site, Vitebsk
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Dinant
  - Research Site, Liège
  - Research Site, Yvoir
- Czechia (5):
  - Research Site, Brno
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Zlín
- France (17):
  - Research Site, Angers
  - Research Site, Argenteuil
  - Research Site, Colombes
  - Research Site, La Roche-sur-Yon
  - Research Site, Le Chesnay
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site 1, Paris
  - Research Site 2, Paris
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Pontoise
  - Research Site, Strasbourg
  - Research Site, Tourcoing
  - Research Site, Tours
- Georgia (3):
  - Research Site 1, Kutaisi
  - Research Site 2, Kutaisi
  - Research Site, Tbilisi
- Greece (4):
  - Research Site 1, Athens
  - Research Site 2, Athens
  - Research Site 1, Larissa
  - Research Site 2, Larissa
- Hungary (5):
  - Research Site 3, Budapest
  - Research Site 2, Budapest
  - Research Site 1, Budapest
  - Research Site, Debrecen
  - Research Site, Nyíregyháza
- Mexico (3):
  - Research Site 1, Guadalajara
  - Research Site 2, Guadalajara
  - Research Site, Monterrey
- Peru (3):
  - Research Site, Lima
  - Research Site, Miraflores
  - Research Site, San Martín de Porres
- Poland (2):
  - Research Site, Opole
  - Research Site, Warsaw
- Russia (10):
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site 2, Novosibirsk
  - Research Site 3, Novosibirsk
  - Research Site 1, Novosibirsk
  - Research Site 2, Saint Petersburg
  - Research Site 3, Saint Petersburg
  - Research Site 4, Saint Petersburg
  - Research Site 1, Saint Petersburg
  - Research Site, Tomsk
- South Korea (7):
  - Research Site 1, Gyeonggi-do
  - Research Site 2, Gyeonggi-do
  - Research Site 2, Seoul
  - Research Site 1, Seoul
  - Research Site 3, Seoul
  - Research Site 4, Seoul
  - Research Site, Wŏnju
- Spain (9):
  - Research Site 1, Barcelona
  - Research Site 2, Barcelona
  - Research Site 3, Barcelona
  - Research Site 4, Barcelona
  - Research Site, Madrid
  - Research Site, Mataró
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Tarragona
- Taiwan (9):
  - Research Site 1, Kaohsiung City
  - Research Site 2, Kaohsiung City
  - Research Site 2, Taichung
  - Research Site 1, Taichung
  - Research Site, Tainan
  - Research Site 1, Taipei
  - Research Site 4, Taipei
  - Research Site 2, Taipei
  - Research Site 3, Taipei
- Ukraine (3):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kiev
  - Research Site, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Matching placebo
  placebo: matching placebo
Period: Overall Study
Arm/Group | AR-105 | Control
Started | 79 (Safety and ITT population) | 79 (Safety and ITT population)
Completed | 49 (Safety and ITT population) | 62 (Safety and ITT population)
Not Completed | 30 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-105 | Control | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.83) | 61.2 (15.58) | 62.3 (14.73)
Age, Customized [Count of Participants; unit: Participants]
  Age </= 64 years | 40 | 39 | 79
  Age > 64 years | 39 | 40 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 62 | 58 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 73 | 74 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Number of participants per Country
  participants
    Hungary | 10 | 8 | 18
    United States | 3 | 4 | 7
    Czechia | 5 | 5 | 10
    Ukraine | 6 | 11 | 17
    Belarus | 7 | 5 | 12
    Russia | 21 | 21 | 42
    Spain | 4 | 3 | 7
    Greece | 5 | 2 | 7
    Belgium | 3 | 3 | 6
    Taiwan | 2 | 3 | 5
    Georgia | 1 | 0 | 1
    France | 10 | 14 | 24
    South Korea | 2 | 0 | 2
World Regions [Count of Participants; unit: Participants] — Actual Regions of Enrollment
  Participants
    Americas | 3 | 4 | 7
    Eastern Europe | 50 | 50 | 100
    Western Europe | 22 | 22 | 44
    Asia | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure on Day 21
Description: A summary of the number (%) of patients who were cured on or before Day 21 (micro-ITT population) is provided, by treatment group
Time Frame: 21 days following dosing
Measure: Count of Participants; unit: Participants
Arm/Group | AR-105 | Control
Number analyzed (Participants) | 70 | 67
Participants
  Observed Cured | 34 | 37
  Imputed Cured | 6 | 5
  Not Cured | 25 | 20
  Reinfection same pathogen | 5 | 2
  New Infection Different Pathogen | 0 | 3
  New infection Unknown pathogen | 0 | 0
Statistical Analysis 1: Comparison: AR-105 vs Control; Test type: Superiority — comparison between the treatment and placebo; p = 0.6154, Cochran-Mantel-Haenszel — P-value was obtained with the stratified CMH test adjusted for baseline randomization strata; Risk Difference (RD) = -5.54, 95% CI 2-sided [-21.9 to 10.8]

2. Secondary Outcome: Clinical Cure on Day 7
Description: A summary of the number (%) of patients who were cured on or before Day 7 (micro-ITT population) is provided, by treatment group
Time Frame: 7 days following dosing
Measure: Count of Participants; unit: Participants
Arm/Group | AR-105 | Control
Number analyzed (Participants) | 70 | 67
Participants
  Cured Observed | 16 | 18
  Cured Imputed | 0 | 0
  Not Cured | 52 | 47
  Re-infection Same Pathogen | 1 | 0
  New Infection Different Pathogen | 1 | 1
  New Infection Unknown Pathogen | 0 | 1
Statistical Analysis 1: Comparison: AR-105 vs Control; Comparison between the treatment and placebo; Test type: Superiority; p = 0.8426, Cochran-Mantel-Haenszel — P-value was obtained with the stratified CMH test adjusted for baseline randomization strata; Risk Difference (RD) = 4.01, 95% CI 2-sided [-18.5 to 10.5]

3. Secondary Outcome: Clinical Cure on Day 14
Description: A summary of the number (%) of patients who were cured on or before Day 14 (micro-ITT population) is provided by treatment group
Time Frame: 14 days following dosing
Measure: Count of Participants; unit: Participants
Arm/Group | AR-105 | Control
Number analyzed (Participants) | 70 | 67
Participants
  Observed Cured | 36 | 31
  Imputed Cured | 1 | 2
  Not Cured | 29 | 30
  Reinfection same pathogen | 1 | 0
  New Infection Different Pathogen | 2 | 4
  New infection Unknown Pathogen | 1 | 0
Statistical Analysis 1: Comparison: AR-105 vs Control; Comparison between the treatment and placebo; Test type: Superiority — comparison between the treatment and placebo; p = 0.3562, Cochran-Mantel-Haenszel — P-value was obtained with the stratified CMH test adjusted for baseline randomization strata; P value CMH = 3.6, 95% CI 2-sided [-13.1 to 20.3]

4. Secondary Outcome: Clinical Cure on Day 28
Description: A summary of the number (%) of patients who were cured on or before Day 28 (micro-ITT population) is provided by treatment group
Time Frame: 28 days following dosing
Measure: Count of Participants; unit: Participants
Arm/Group | AR-105 | Control
Number analyzed (Participants) | 70 | 67
Participants
  Observed Cured | 35 | 38
  Imputed Cured | 9 | 6
  Not Cured | 23 | 16
  Reinfection same pathogen | 3 | 3
  New Infection Different Pathogen | 0 | 4
  New infection Unknown Pathogen | 0 | 0
Statistical Analysis 1: Comparison: AR-105 vs Control; Test type: Superiority — Comparison between the treatment and placebo; p = 0.8472, Cochran-Mantel-Haenszel — P-value was obtained with the stratified CMH test adjusted for baseline randomization strata; P value CMH = -2.81, 95% CI 2-sided [-18.9 to 13.2]

5. Post Hoc Outcome: Absolute Difference Clinical Cure at Day 14 and 21 for Study 1
Description: Difference in percentage of clinical cure rates between the two treatment groups
Time Frame: Up to Day 21
Measure: Count of Participants; unit: Participants
Groups:
- Subset AR-105 Study1; Subset Placebo Study1: Using the appropriate clinical severity, level of CRP and adequate antibiotic criteria, patients were subdivided into subgroups to identify a pattern in the clinical cure rates in both treatment groups. The results suggest the presence of heterogeneity of factors influencing the clinical cure rates, where only a quite small sample is evaluable. A subset of patients had the following characteristics and were found to belong to
  1. appropriate clinical Severity
  2. inadequate antibiotic regimen and
  3. lower 3rd quartile of level of CRP
Arm/Group | Subset AR-105 Study1 | Subset Placebo Study1
Number analyzed (Participants) | 9 | 18
Participants
  Cured Day 14 | 6 | 8
  Cured Day 21 | 7 | 10
Statistical Analysis 1: Comparison: Subset AR-105 Study1 vs Subset Placebo Study1; Data for Day 14; Test type: Superiority; p = 0.4616, Chi-squared — Marginally statistically significant only if p<0.1; Mean Difference (Final Values) = 22.3, 95% CI 2-sided [-16.2 to 60.6]
Statistical Analysis 2: Comparison: Subset AR-105 Study1 vs Subset Placebo Study1; Data for Day 21; Test type: Superiority; p = 0.4053, Chi-squared — Data for Day 21; Mean Difference (Final Values) = 22.3, 95% CI 2-sided [-13.3 to 57.8]

6. Post Hoc Outcome: Absolute Difference Clinical Cure at Day 14 and 21 for Study 2
Description: Difference in percentage of clinical cure rates between the two treatment groups
Time Frame: Up to Day 21
Measure: Count of Participants; unit: Participants
Groups:
- Subset AR-105 Study2; Subset Placebo Study2: Using the appropriate clinical severity, level of CRP and adequate antibiotic criteria, patients were subdivided into subgroups to identify a pattern in the clinical cure rates in both treatment groups. The results suggest the presence of heterogeneity of factors influencing the clinical cure rates, where only a quite small sample is evaluable. A subset of patients had the following characteristics and were found to belong to
  1. appropriate clinical Severity
  2. inadequate antibiotic regimen and
  3. lower 3rd quartile of level of CRP
Arm/Group | Subset AR-105 Study2 | Subset Placebo Study2
Number analyzed (Participants) | 3 | 7
Participants
  Cured Day 14 | 2 | 2
  Cured Day 21 | 2 | 3
Statistical Analysis 1: Comparison: Subset AR-105 Study2 vs Subset Placebo Study2; Data for Day 14; Test type: Superiority; p = 0.0833, Chi-squared — Marginally statistically significant only if p<0.1; Mean Difference (Final Values) = 38.1, 90% CI 2-sided [-14.8 to 90.9]
Statistical Analysis 2: Comparison: Subset AR-105 Study2 vs Subset Placebo Study2; Data for Day 21; Test type: Superiority; p = 0.5151, Chi-squared — Data for Day 21; Marginally statistically significant only if p<0.1 Day 21; Mean Difference (Net) = 23.8, 90% CI 2-sided [-30.5 to 78.1]

ADVERSE EVENTS:
Time Frame: 1 month: from administration day (Day 0) up to Day 28 (28 days after administration)
Arm/Group | AR-105 | Control
All-Cause Mortality (participants affected / at risk) | 25/79 | 13/79
Serious Adverse Events (participants affected / at risk) | 36/79 | 22/79
Other Adverse Events (participants affected / at risk) | 73/79 | 73/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-105 (N=79) | Control (N=79)
Circulatory Collapse (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 7 | 4
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 3 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Rhythm idioventricular (Cardiac disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Brain oedema (Nervous system disorders) | 3 | 0
Coma (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 5 | 3
Systemic candida (Infections and infestations) | 0 | 1
Arterial rupture (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-105 (N=79) | Control (N=79)
Hypotension (Vascular disorders) | 14 | 9
Multiple organ dysfunction syndrome (General disorders) | 10 | 4
Oedema peripheral (General disorders) | 1 | 4
Pyrexia (General disorders) | 5 | 3
Agitation (Nervous system disorders) | 4 | 2
Alanine aminotransferase increased (Investigations) | 0 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 6
Atrial fibrillation (Cardiac disorders) | 6 | 7
Bradycardia (Cardiac disorders) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 16 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Brain oedema (Nervous system disorders) | 5 | 0
Delirium (Nervous system disorders) | 4 | 2
Insomnia (Nervous system disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 13
Nausea (Gastrointestinal disorders) | 3 | 4
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 6
Hypovolaemia (Metabolism and nutrition disorders) | 4 | 3
Cystitis (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 5 | 5
Sepsis (Infections and infestations) | 5 | 0
Septic shock (Infections and infestations) | 6 | 5
Tracheobronchitis (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 1 | 6

LIMITATIONS AND CAVEATS:
A post-hoc analysis was performed on the data reviewed by the AC, using the appropriate clinical severity, adequate antibiotic criteria and the inflammatory status of the patient (level of C-reactive protein [CRP]).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03027609/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03027609/SAP_001.pdf